CLINICAL TRIAL: NCT04800549
Title: The Effect of Black Mulberry Lollipop and Sodium Bicarbonate Used in Oral Care on Prevention of Oral Mucositis Among Children Receiving Chemotherapy Due to Cancer
Brief Title: Effect of Black Mulberry Lollipop on Prevention of Oral Mucositis in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sapanca Ilce Devlet Hastanesi (Other Government)
Collaborators: Okan University (Other)
Responsible Party: Principal Investigator, ebru kaya, Principal Investigator, Sapanca Ilce Devlet Hastanesi
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: SapancaH
Record Dates: First submitted 2019-12-13; First posted 2021-03-16 (Actual); Last update posted 2021-03-16 (Actual); Status verified 2021-03

CONDITIONS: Oral Mucositis
Keywords: Keywords: chemotherapy, oral mucositis, black mulberry, bicarbonate, paediatric oncology
MeSH Terms: conditions — Stomatitis

STUDY DESIGN:
Intervention Model Description: The power of the test in the study was calculated by using G*Power 3.1 program. While Type I error is 0.05 and the power of the test is 0.80 (α= 0.05, 1-β= 0.80), minimal sample size was calculated as 62 children (31 children in each group). By considering the losses that may occur from the sample during the study due to any reason, it was planned to include 40 children in both experimental and control groups. Follow-up lost occurred in 5 patients from experimental group and 6 patients in the control group during the study. The study was completed with 69 paediatric patients including 34 in the experimental group and 35 in the control group.
Masking Description: The power of the test in the study was calculated by using G*Power 3.1 program. While Type I error is 0.05 and the power of the test is 0.80 (α= 0.05, 1-β= 0.80), minimal sample size was calculated as 62 children (31 children in each group). By considering the losses that may occur from the sample during the study due to any reason, it was planned to include 40 children in both experimental and control groups. Follow-up lost occurred in 5 patients from experimental group and 6 patients in the control group during the study. The study was completed with 69 paediatric patients including 34 in the experimental group and 35 in the control group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- METHOD (Experimental): The power of the test in the study was calculated by using G*Power 3.1 program. While Type I error is 0.05 and the power of the test is 0.80 (α= 0.05, 1-β= 0.80), minimal sample size was calculated as 62 children (31 children in each group). By considering the losses that may occur from the sample during the study due to any reason, it was planned to include 40 children in both experimental and control groups. Follow-up lost occurred in 5 patients from experimental group and 6 patients in the control group during the study. The study was completed with 69 paediatric patients including 34 in the experimental group and 35 in the control group.
  Interventions: Other: Oral Mucositis

INTERVENTIONS:
Other: Oral Mucositis — The data of the study were obtained by conducting six interviews with each child and the family. The first interview was conducted before starting to treatment on the first day of the treatment, the second interview was conducted on the 2nd day after the treatment and the following interviews were conducted on the 4th, 8th, 16th, and 21st days and in-mouth mucosa of the patient was evaluated by taking in-mouth pictures following interviewing with the child and the family. Oral care application was conducted four times a day with sodium bicarbonate solution and a lollipop made with black mulberry syrup (after meals and before going to the bed at night). Oral care was first conducted by the researcher, the oral care was then taught to the patient and patient's relatives and the application was evaluated. Figure 1 shows the study design.

SUMMARY:
THE EFFECT OF BLACK MULBERRY LOLLIPOP AND SODIUM BICARBONATE USED IN ORAL CARE ON PREVENTION OF ORAL MUCOSITIS AMONG CHILDREN RECEIVING CHEMOTHERAPY DUE TO CANCER

DETAILED DESCRIPTION:
The study was conducted experimentally to determine the effect of black mulberry lollipop and sodium bicarbonate used in oral care on prevention of oral mucositis in children followed up due to the diagnosis of cancer. Sodium bicarbonate and black mulberry treatment were compared to prevent oral mucositis in 69 children receiving chemotherapy due to cancer. While 35 children were assigned to the experimental group (sodium bicarbonate + black mulberry lollipop application), 34 were assigned to the control group (sodium bicarbonate application).

ELIGIBILITY:
Inclusion Criteria:

* Being in the age group of 3-18 years
* Being hospitalised for chemotherapy treatment
* Not having oral mucositis
* No using another method to protect oral mucosa during the study period
* Not having the history of black mulberry (similar fruit berries, blackberries, etc.) allergy
* Not having intolerance to cold

Exclusion Criteria:

-Not having food in mouth

Ages: 3 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 69 (Actual)
Dates: Start 2016-02 (Actual); Primary Completion 2017-02 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
Patient Follow-up Form | 3 minute
  It has 16 questions prepared by the researcher utilising literature and including sociodemographic characteristic and oral care habits of the child and family.
Children's International Mucositis Evaluation Scale | 2 minute
  Tomlison et al. (2010) developed Children's International Mucositis Evaluation Scale (ChIMES) in order to evaluate the difficulty experienced by children with cancer due to mouth/throat pain developing depending on mucositis. Yavuz et al., (2011) conducted the validity and reliability study of the Turkish version of the scale. The scale consists of six (6) questions and it is an easy-to-apply form that can be answered with the child's facial expressions.
Nurse Observation Chart of Child Mucositis Evaluation | 10 minute
  It was prepared in parallel with Oral Mucositis Evaluation Index of the World Health Organization and formed to monitor formation or level of oral mucositis in children on the first, second, fourth, eights, sixteenth and twenty first days.

CONTACTS AND LOCATIONS:
Locations (1):
- Sağlık Bakanlığı Sapanca Ilçe Hastanesi, Sakarya, Türkiye, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided